CLINICAL TRIAL: NCT04819321
Title: Study of White Adipose Tissue Remodeling by Cryolipolysis in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Allergan Sales, LLC (Industry)
Responsible Party: Principal Investigator, Adaliene Versiani M. Ferreira, Adaliene Versiani M. Ferreira, PHD, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 30339520.8.0000.5149
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Lipid Metabolism Disorders; Metabolic Disease
Keywords: CoolSculpting; adipose tissue; cryolipolysis; browning
MeSH Terms: conditions — Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: The sample will comprise 12 adult women (aged 18 to 40 years) and overweight (BMI> 24.9 kg / m² and <30.0 kg / m²).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CoolSculpting® System (Experimental): A treatment is comprised of timed segments of cooling and heating; a vacuum treatment may include an optional massage
  Interventions: Device: CoolSculpting® System

INTERVENTIONS:
Device: CoolSculpting® System — A treatment is comprised of timed segments of cooling and heating; a vacuum treatment may include an optional massage

SUMMARY:
The sample will comprise 12 adult women (aged 18 to 40 years) and overweight (BMI> 24.9 kg / m² and <30.0 kg / m²). The experimental design will consist of four assessments. In the first assessments a structured questionnaire will be applied to obtain health and food consumption data, in addition to evaluate anthropometric (weight, height, waist and hip circumference), and collection of blood. In addition, an ultrasound examination, digital photography and biopsy of the subcutaneous WAT, of the abdominal region, will be performed. After 30 day subjects will undergo CoolSculpting treatment(s) in an outpatient clinical setting. The treatment is comprised of timed segments of cooling and heating; a vacuum treatment may include an optional massage. Treatments will be administered according to the User Manual CoolSculpting System. The volunteers will return for the biopsy of the subcutaneous WAT, from the abdominal region, in 3 days after the procedure. In 4º assessment, 60 days after cryolipolysis, all evaluations performed in the first assessment will be repeated and to evaluate overall patient satisfaction for non-invasive fat reduction in CoolSculpting subjects.

DETAILED DESCRIPTION:
This is a longitudinal, non-randomized clinical trial to assess the biology of AT after the use of cryolipolysis. The study will be developed at "Clinica Dra Ligia Colucci" in partnership with the Federal University of Minas Gerais (UFMG). The project will be submitted for evaluation by the Research Ethics Committee (COEP / UFMG). All participants must sign the informed consent form (ICF), before the study begins.

The experimental design will consist of five stages. Initially, women will be public recruitment. Through telephone contact, the inclusion and exclusion criteria will be verified, and volunteers who meet the criteria will be invited to attend the clinic for the first stage of the study. The presentation of the research, will be carried out 7 days before the beginning of the treatment, will consist of presenting the project to the volunteers, explaining all the risks and benefits related to the study and request the signature of the ICF. After 7 days, the volunteers must return to the clinic, then start the study. In the initial evaluation, an anamnesis of the volunteers will be carried out with a standardized form, including socioeconomic and clinical data, data on the use of medications, alcohol consumption, physical activity and food consumption. In addition, anthropometric assessments will be performed where weight, height, waist, abdominal and hip circumference will be measured. Ultrasonography will also be performed; the abdominal region will be photographed and blood will be collected to measure lipolytic and inflammatory markers and a biopsy of the subcutaneous WAT in the lower abdomen via umbilical scar. In addition, questionnaires will be applied to check the volunteers' satisfaction with the treatment. After 30 days, the volunteers must return to the clinic for time 0 (T0), where anthropometric assessments will be repeated as control variables. Ultrasound and blood collection will also be performed. Then the volunteers will be submitted to cryolipolysis in the abdominal region by the Coolsculpting® system. After 3 days of performing the Coolsculpting® procedure, the volunteers must return to the clinic for time 3 (T3), to perform a new biopsy of the subcutaneous WAT in the lower abdomen via the umbilical scar. After 60 days of the cryolipolysis, the volunteers must return to the clinic for the time 60 (T60), where all the evaluations of the initial evaluation will be carried out again and a personal satisfaction questionnaire will be applied in relation to the result of the procedure. Therefore, the study will total 97 days of monitoring of women, who will be instructed to maintain healthy lifestyle habits, according to the conventional lifestyle of each one of them. The data, images and biological materials (blood and adipose tissue biopsy) collected in the research will be filed with the researcher responsible for a period of 5 (five) years at the Experimental Nutrition Laboratory, room 315, of the UFMG School of Nursing and after that time will be destroyed. In case of occurrence of paradoxical adipose hyperplasia after the procedure, a case study of the possible affected patients will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Subject has clearly visible fat in the flanks and/or abdomen, which in the investigator's opinion, may benefit from the treatment.

Subject has not had weight change fluctuations exceeding 4.5 kg (or 5% of body weight) in the preceding month.

Subject has a BMI of 24.9 to 30. A BMI is defined as weight in kilograms divided by height in meters squared (kg/m2).

Subject agrees to maintain weight (ie, within 5% of body weight) by not making any changes in diet or exercise routine during the course of the study.

Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

Exclusion Criteria:

* Subject has had liposuction, or another surgical procedure(s) or mesotherapy in area of intended treatment.

Subject has had a non-invasive fat reduction and/or body contouring procedure in the area(s) of intended treatment within the past 12 months.

Subject needs to administer, or has a known history of subcutaneous injections into the area(s) of intended treatment (eg, cortisone, heparin, insulin) within the past 6 months.

Subject is pregnant or intending to become pregnant. Subject is lactating or has been lactating in the past 6-9 months. Subject is unable or unwilling to comply with study requirements. Subject is currently enrolled in a clinical study of any unapproved investigational device, investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.

Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system or any other metal containing implant.

Subject with known history of cryoglobulinemia, cold agglutinin disease, or paroxysmal cold hemoglobinuria.

Subject with known sensitivity to cold or has any condition with a known response to cold exposure that limits blood flow to the skin such as cold urticaria or Raynaud's disease, or Chilblains (pernio).

Subject with known sensitivity or allergy to fructose, glycerin, isopropyl alcohol, or propylene glycol.

Subject with impaired peripheral circulation in the area to be treated Subject with neuropathic disorders such as post-herpetic neuralgia or diabetic neuropathy.

Subject with impaired skin sensation. Subject with open or infected wounds. Subject with bleeding disorders, or concomitant use of blood thinners, or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.

Subject with recent surgery or scar tissue in the area to be treated. Subject has history of hernia in or adjacent to the treatment area(s) site. Subject with skin conditions such as eczema, dermatitis, or rashes in the area to be treated.

Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).

Subject is taking or has taken diet pills or supplements within the past 6 months.

Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Subject diagnosed with fibrosis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue biology | 3 days after the procedure
  Fat cell death after cooling by cryolipolysis
Change in volume of fat from baseline | 60 days after the procedure
  To evaluate change in volume of fat after CoolSculpting treatment(s) using ultrasound and photography.

SECONDARY OUTCOMES:
Decrease in abdominal circumference | 60 days after the procedure
  decreased abdominal circumference after death of adipocytes
Browning of white adipose tissue | 3 days after the procedure
  browning of white adipose tissue

OTHER OUTCOMES:
Paradoxical adipose hyperplasia | Up to 60 days after the procedure
  In case of occurrence of paradoxical adipose hyperplasia after the procedure, a case study of the possible affected patients will be carried out

CONTACTS AND LOCATIONS:
Overall Officials: Mariele L Silva, Master, Study Chair — Federal University of Minas Gerais; Amanda CC Oliveira, Master, Study Chair — Federal University of Minas Gerais; Adma M Babetto, Student, Study Chair — Federal University of Minas Gerais; Adaliene VM Ferreira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Departamento de Nutrição Escola de Enfermagem Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal M, Kern PA, Nikolajczyk BS. The Immune System in Obesity: Developing Paradigms Amidst Inconvenient Truths. Curr Diab Rep. 2017 Aug 15;17(10):87. doi: 10.1007/s11892-017-0917-9. PMID 28812211
- [Background] Aldiss P, Betts J, Sale C, Pope M, Budge H, Symonds ME. Exercise-induced 'browning' of adipose tissues. Metabolism. 2018 Apr;81:63-70. doi: 10.1016/j.metabol.2017.11.009. Epub 2017 Nov 16. PMID 29155135
- [Background] Avram MM, Harry RS. Cryolipolysis for subcutaneous fat layer reduction. Lasers Surg Med. 2009 Dec;41(10):703-8. doi: 10.1002/lsm.20864. PMID 20014262
- [Background] Garibyan L, Sipprell WH 3rd, Jalian HR, Sakamoto FH, Avram M, Anderson RR. Three-dimensional volumetric quantification of fat loss following cryolipolysis. Lasers Surg Med. 2014 Feb;46(2):75-80. doi: 10.1002/lsm.22207. Epub 2013 Dec 3. PMID 24535759
- [Background] Harms M, Seale P. Brown and beige fat: development, function and therapeutic potential. Nat Med. 2013 Oct;19(10):1252-63. doi: 10.1038/nm.3361. Epub 2013 Sep 29. PMID 24100998
- [Background] Ingargiola MJ, Motakef S, Chung MT, Vasconez HC, Sasaki GH. Cryolipolysis for fat reduction and body contouring: safety and efficacy of current treatment paradigms. Plast Reconstr Surg. 2015 Jun;135(6):1581-1590. doi: 10.1097/PRS.0000000000001236. PMID 26017594
- [Background] Kajimura S, Spiegelman BM, Seale P. Brown and Beige Fat: Physiological Roles beyond Heat Generation. Cell Metab. 2015 Oct 6;22(4):546-59. doi: 10.1016/j.cmet.2015.09.007. PMID 26445512
- [Background] Kilmer SL. Prototype CoolCup cryolipolysis applicator with over 40% reduced treatment time demonstrates equivalent safety and efficacy with greater patient preference. Lasers Surg Med. 2017 Jan;49(1):63-68. doi: 10.1002/lsm.22550. Epub 2016 Jun 21. PMID 27327898
- [Background] Kilmer SL, Burns AJ, Zelickson BD. Safety and efficacy of cryolipolysis for non-invasive reduction of submental fat. Lasers Surg Med. 2016 Jan;48(1):3-13. doi: 10.1002/lsm.22440. Epub 2015 Nov 26. PMID 26607045
- [Background] Krueger N, Mai SV, Luebberding S, Sadick NS. Cryolipolysis for noninvasive body contouring: clinical efficacy and patient satisfaction. Clin Cosmet Investig Dermatol. 2014 Jun 26;7:201-5. doi: 10.2147/CCID.S44371. eCollection 2014. PMID 25061326
- [Background] Lee P, Smith S, Linderman J, Courville AB, Brychta RJ, Dieckmann W, Werner CD, Chen KY, Celi FS. Temperature-acclimated brown adipose tissue modulates insulin sensitivity in humans. Diabetes. 2014 Nov;63(11):3686-98. doi: 10.2337/db14-0513. Epub 2014 Jun 22. PMID 24954193
- [Background] Manstein D, Laubach H, Watanabe K, Farinelli W, Zurakowski D, Anderson RR. Selective cryolysis: a novel method of non-invasive fat removal. Lasers Surg Med. 2008 Nov;40(9):595-604. doi: 10.1002/lsm.20719. PMID 18951424
- [Background] Nelson AA, Wasserman D, Avram MM. Cryolipolysis for reduction of excess adipose tissue. Semin Cutan Med Surg. 2009 Dec;28(4):244-9. doi: 10.1016/j.sder.2009.11.004. PMID 20123423
- [Background] Shek SY, Chan NP, Chan HH. Non-invasive cryolipolysis for body contouring in Chinese--a first commercial experience. Lasers Surg Med. 2012 Feb;44(2):125-30. doi: 10.1002/lsm.21145. PMID 22334296
- [Background] Leal Silva H, Carmona Hernandez E, Grijalva Vazquez M, Leal Delgado S, Perez Blanco A. Noninvasive submental fat reduction using colder cryolipolysis. J Cosmet Dermatol. 2017 Dec;16(4):460-465. doi: 10.1111/jocd.12383. Epub 2017 Sep 12. PMID 28901051
- [Background] Stevens WG, Bachelor EP. Cryolipolysis conformable-surface applicator for nonsurgical fat reduction in lateral thighs. Aesthet Surg J. 2015 Jan;35(1):66-71. doi: 10.1093/asj/sju024. PMID 25568236
- [Background] Sun K, Kusminski CM, Scherer PE. Adipose tissue remodeling and obesity. J Clin Invest. 2011 Jun;121(6):2094-101. doi: 10.1172/JCI45887. Epub 2011 Jun 1. PMID 21633177
- [Background] Yoneshiro T, Aita S, Matsushita M, Kayahara T, Kameya T, Kawai Y, Iwanaga T, Saito M. Recruited brown adipose tissue as an antiobesity agent in humans. J Clin Invest. 2013 Aug;123(8):3404-8. doi: 10.1172/JCI67803. Epub 2013 Jul 15. PMID 23867622